CLINICAL TRIAL: NCT00064896
Title: Technical Development of Interventional Cardiovascular Magnetic Resonance Imaging
Brief Title: Technical Development of Cardiovascular Magnetic Resonance Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030250; 03-H-0250
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10-26

CONDITIONS: Peripheral Artery Disease
Keywords: Blood Flow; Revascularization; Image Fusion; Fluoroscopy; MRI; Chronic Total Occlusion of Arteries; Claudication; Safety; Atherosclerosis; Cardiovascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Atherosclerosis; Cardiovascular Diseases

INTERVENTIONS:
Procedure: MRI

SUMMARY:
The goal of this study is to develop advances in cardiovascular diagnostic and treatment methods using magnetic resonance imaging (MRI), a test that uses a strong magnetic field and radio waves to show anatomic detail. For the scan, the patient lies on a table in a cylinder containing a magnetic field. He or she can communicate with a staff member at all times during the procedure.

Patients 18 years of age or older who require 1) catheterization of the leg arteries for diagnosis or treatment of blocked arteries, or 2) heart catheterization for diagnosis or treatment of coronary artery disease or other heart problems may be eligible for this study. Participants will undergo one of the following procedures:

Blood Flow Measurement Using Standard Techniques and MRI

For patients with blockage in a leg artery, blood flow will be measured before and after successful catheter-based treatment (angioplasty or stenting) using standard venous occlusion plethysmography and a newer MRI technique. (Patients whose treatment is not successful will not undergo follow-up blood flow measurements in this study.) For venous occlusion plethysmography, a large pressure cuff is placed around the upper or lower legs. Thin elastic bands called a strain gauge are placed around the calves to measure blood blow to the legs. The pressure cuffs are inflated for 5 minutes, preventing blood from flowing to the legs, and are then deflated, allowing the blood to rush to the legs. A smaller cuff is inflated to a low pressure, and the strain gauge measures this maximum blood flow to the legs for 1 or 2 more minutes. For the new MRI technique, blood flow is measured while the patient is in the MRI scanner. Flow is first measured with the patient at rest. Then, the large pressure cuff is inflated for 5 minutes. The cuff is deflated and additional images are taken. Before the cuff is deflated, a dye called gadolinium contrast is injected into an arm vein to brighten the images. Patients may undergo six to eight cuff inflations on four to six different days.

Fusion of X-Ray and MRI Images of Peripheral Arteries

For patients with blockage in a leg artery Participants will undergo catheterization and MRI of the legs. Special plastic beads are taped to the leg(s) to help compare the MRI and x-ray pictures. For the catheterization procedure, x-rays of the blood vessels are taken to guide placement of the catheters. Contrast dye is injected to brighten the images of the blood vessels. These injections work well in normal and partly blocked arteries, but not in arteries that are completely blocked. For this study, patients first have an MRI scan of their legs. During the scan, gadolinium contrast dye is injected into an arm vein. Then, during the catheterization procedure, a computer aligns the MRI pictures with the x-ray pictures to see if the combined images allow the doctor to better see where to place the catheters.

Fusion of X-ray and MRI Images of the Heart

For patients undergoing heart catheterization will undergo MRI and heart catheterization. Special plastic beads are taped to the chest to help compare the MRI and x-ray pictures. Patients first have an MRI scan of their heart. During the scan, gadolinium contrast dye is injected into an arm vein. Then, during the catheterization procedure, a computer aligns the MRI pictures with the x-ray pictures to see if the combined images allow the doctor to learn more about the pattern of heart disease.

Heart rhythm, blood pressure, heart function, and breathing will be monitored during all the MRIs.

DETAILED DESCRIPTION:
Cardiovascular interventional procedures are minimally-invasive, catheter-based treatments such as coronary artery angioplasty and stenting. These procedures generally can be conducted on awake patients with few complications, and were developed as alternatives to conventional open surgery. Conventional cardiovascular interventional procedures are conducted by physicians manipulating medical devices inside patients under the guidance of fluoroscopic x-ray.

We are developing minimally-invasive cardiovascular interventional procedures using real-time magnetic resonance imaging, also known as MR Fluoroscopy. These procedures have the advantage of excellent imaging without surgery and without radiation exposure or toxic contrast agents (dyes). Moreover, because MR Fluoroscopy can produce excellent images of soft tissue, blood, and of three-dimensional structures, it may be possible to guide minimally-invasive procedures not possible even with invasive surgery.

The goal of this protocol is to develop and test incremental technical advances in patients.

ELIGIBILITY:
* INCLUSION CRITERIA FOR ALL ARMS OF THE PROTOCOL:

Subjects with known or suspected cardiovascular disease will be eligible for participation in this protocol. The subject is eligible under the following conditions:

Subject's age is greater than 18 years of age.

Expected to undergo, or having undergone, a clinically-indicated diagnostic or therapeutic catheterization procedure or MRI angiogram procedure.

Additional Inclusion Criteria for Section #4: Magnetic Resonance Imaging of Peripheral Arterial Atherosclerosis

-Known or suspected peripheral artery occlusion.

EXCLUSION CRITERIA FOR ALL ARMS OF THE PROTOCOL:

Subjects with absolute contraindications to MRI scanning will be excluded. These contraindications include subjects with the following devices:

* Implanted cardiac pacemaker or defibrillator
* Central nervous system aneurysm clips
* Implanted neural stimulator
* Cochlear implant
* Ocular foreign body (e.g. metal shavings)
* Insulin pump
* Metal shrapnel or bullet.

When subjects can provide evidence that their implanted device is labeled compatible with MRI, exceptions to the above exclusions can be made and recorded in the note. Furthermore, the FOLLOWING SUBJECT GROUPS WILL BE EXCLUDED because of the administration of MRI CONTRAST AGENTS:

* Pregnant women (Subjects who are uncertain as to whether they are pregnant will be required to have a screening urine or blood pregnancy test) or Lactating Women.
* Subjects with hemoglobinopathies
* Subjects with renal disease (eGFR[R] less than 30 mL/min/1.73m(2))

Glomerular filtration rate will be estimated using the MDRD 2005 revised study formula:

eGFR (mL/min/1.73m (2)) equal 175 x (standardized Scr) (-1.154) x (age) (-0.203) x 0.742 (if the subject is female) or x 1.212 (if the subject is black)

However, if the eGFR less than 30 mL/min/1.73m(2) and gadolinium contrast exposure is thought likely to reduce the overall risk of the medically necessary interventional procedure in Specific Aim number 2, then with informed consent and the concurrence of the attending physician, the patient may be enrolled in the study. This would be documented in the medical record, and the IRB would be notified.

Additional Exclusion Criteria for Section #2: Lower Extremity Perfusion Measures

A patent autologous or prosthetic bypass graft that would require compression during arterial occlusion to induce reactive hyperemia. This exclusion is intended to avoid graft injury and possible thrombosis. If an old graft is known to be non-functional, from radiocontrast or MRI angiography, then this exclusion does not apply.

A patent intravascular stent in a territory that would be compressed during arterial occlusion to induce reactive hyperemia. This exclusion is intended to avoid theoretical stent crush or fracture. If the stented vessel is known to be completely occluded, from radiocontrast or MRI angiography, then this exclusion does not apply. However, occlusive cuffs may be placed above or below stent devices to avoid this theoretical complication.

Active deep vein thrombosis of the lower extremity based on clinical findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-07-14; Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
To develop, test, and provide adjunctive information to the operator derived from MRI during the management of patients being considered for, or undergoing, invasive procedures.

SECONDARY OUTCOMES:
This protocol aims to develop and test novel MRI techniques in patients being treated for cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Murphy KP, Szopinski KT, Cohan RH, Mermillod B, Ellis JH. Occurrence of adverse reactions to gadolinium-based contrast material and management of patients at increased risk: a survey of the American Society of Neuroradiology Fellowship Directors. Acad Radiol. 1999 Nov;6(11):656-64. doi: 10.1016/S1076-6332(99)80114-7. PMID 10894068